CLINICAL TRIAL: NCT01880086
Title: Clomiphene Citrate for the Treatment of Opioid-Induced Androgen Deficiency: Randomized Controlled Clinical Trial
Brief Title: Clomiphene Citrate for the Treatment of Low Testosterone Associated With Chronic Opioid Pain Medication Administration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cornell-1301013472
Record Dates: First submitted 2013-06-07; First posted 2013-06-18 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Hypogonadism; Opioid-Related Disorders; Male Infertility
Keywords: Chronic pain; Low testosterone; Hypogonadism; Opioid analgesics; Narcotics; Opioid-induced androgen deficiency; OPIAD; Male infertility; Clomiphene citrate; Selective Estrogen Receptor Modulators; Testosterone replacement therapy
MeSH Terms: conditions — Hypogonadism; Opioid-Related Disorders; Infertility, Male; Chronic Pain | interventions — Clomiphene; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clomiphene citrate (Experimental): The initial dose of clomiphene citrate will be 25 mg (po, pill by mouth) every other day. This will be started at visit 2, week 0 of the study following diagnosis of low baseline testosterone (serum total testosterone <350 ng/dl in men <55 years, <300 ng/dl in men 55-65 years). Clomiphene citrate dose will be titrated up to a maximum of 50 mg daily according to serum total testosterone levels measured at follow-up visits during the 3 month duration of the study.
  Interventions: Drug: Clomiphene citrate
- Placebo (Placebo Comparator): Placebo pill will be administered (po, pill by mouth) every other day starting at week 0 of the study in men diagnosed with low testosterone. Treatment will be delayed in these men until the 3 month completion of the study, at which time this group may also receive testosterone replacement therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clomiphene citrate
  Other Names: Clomid; Milophene; Serophene
  Arms: Clomiphene citrate
Drug: Placebo — Placebo pill that will have appearance identical to the treatment pill but will not contain active medication.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this randomized controlled clinical trial is to evaluate the effects of clomiphene citrate compared to placebo (substance without active medication) in men who are taking pain medication (opioids) for chronic pain conditions and who have low blood testosterone levels.

The condition of men having low testosterone with long-term pain medication (opioid) usage is called opioid-induced androgen deficiency (OPIAD). Low testosterone can be caused by pain medication effects on part of the brain (hypothalamic-pituitary axis) which ultimately result in decreased testosterone production by the testes. Typical symptoms of low testosterone (hypogonadism) may include decreased muscle mass, increased fat, osteoporosis, anemia, erectile dysfunction, delayed ejaculation. In addition, men with low testosterone may experience decreased attention, and decreased libido, fatigue, and depressed mood. Few studies have looked at hormonal changes caused by long-term opioid usage in men.

Clomiphene citrate, a selective estrogen receptor modulator (SERM) oral medication which inhibits estrogen effects (feedback) on the brain, has been identified by prior studies to raise testosterone in men with low testosterone (due to reasons other than chronic pain medication). Clomiphene citrate is also known to lead to increased sperm production in men with low testosterone unlike testosterone topical or injection medications. Although clomiphene citrate has been studied in hypogonadal men with beneficial outcomes and minimal side effects, no group has previously studied clomiphene citrate as treatment in patients with OPIAD.

DETAILED DESCRIPTION:
Chronic nonmalignant pain is a widespread issue affecting 15-30% of the population. Many patients with chronic pain are responsive to first-line combination of physical modalities and non-opioid analgesics. Up to 20% of these patients, however, require opioid therapy for adequate pain relief. The use of long-acting opioids, including morphine sulfate, oxycodone, fentanyl, and methadone, although effective for pain control, carries risks of addiction, tolerance, and systemic side effects including nausea, itching, constipation, and hypogonadotropic hypogonadism with consequent testosterone depletion (in up to 86% of patients taking chronic pain medication) leading to the multiple adverse effects. Opioid-induced androgen deficiency (OPIAD), occurs with high frequency and persistence, and commonly remains undiagnosed in the pain clinic. Low testosterone may be treated using exogenous testosterone (topical or gel) or other medications such as selective estrogen receptor modulators (i.e. clomiphene citrate). While both medication types increase serum testosterone levels, clomiphene citrate is known to benefit sperm parameters in hypogonadal men while exogenous testosterone is known to inhibit sperm production. Few studies have examined the hormonal changes caused by long-term opioid usage in men, and no studies have formally studied clomiphene citrate for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 years to 65 years
* Low testosterone as defined by criteria (serum total testosterone <350 ng/dl in men <55 years, <300 ng/dl in men 55-65 years)
* EITHER taking opioid pain medication (see A below) OR planning to start new pain medication regimen (see B below)
* A) EITHER continuous opioid treatment for chronic nonmalignant pain for >=6 months receiving one of several specified opioid regimens for the past 1 month (including >=20 mg/day of oral methadone, >=30 mg/day of oral sustained release oxycodone, >=30 mg/day of oral morphine sulfate, >=6 mg/day of oral dilaudid or >= 8 mg/day of dilaudid ER, or >=25 mcg/hr of transdermal fentanyl or buprenorphine, or intrathecal morphine pump)
* B) OR the pain management physician is planning to start pain medication (opioid or non-opioid pain therapy) but you have not received it yet. If this is the case, your testosterone will be checked before starting and during 1 month of pain therapy to determine if you have low testosterone to qualify to begin medication (clomiphene or placebo) treatment in this study.
* BMI (20-35 kg/m2)
* Presence of clear secondary hypogonadism with hypogonadal symptoms and low total testosterone level (confirmed with morning testosterone level <= 350 ng/dL for men age >= 55 and <= 300ng/dl for men age 55-65) or total testosterone <=200 ng/dl (regardless of symptoms). Additionally luteinizing hormone (LH) should be <15 mIU (milli-International unit )/mL (at baseline only). Symptoms of hypogonadism include fatigue, decreased energy level/endurance, depressed mood, decreased libido, erectile dysfunction.
* Chronic nonmalignant pain etiology includes rheumatoid arthritis, osteoarthritis, spinal stenosis, polymyalgia, complex region pain syndrome I and II, neurinoma, phantom limb pain, neuropathic pain of other origin, scoliosis, neck pain, failed back surgery, or chronic pancreatitis.
* All patients must have ability to complete the study in compliance with the protocol, and the ability to understand and provide written informed consent.

Exclusion Criteria:

* Chronic pain of malignant etiology (cancer-related)
* Preexisting testosterone deficiency
* Concomitant use of medication that could interfere with testosterone levels including antidepressant medication, spironolactone, cimetidine, clomiphene (use in the past 1 year), human chorionic gonadotropin (hCG), androgen, estrogen, anabolic steroid, 5-alpha-reductase inhibitors such as finasteride, dehydroepiandrosterone (DHEA), testosterone therapy (topical testosterone within 7 days of study, injectable testosterone within 6 months of study),
* Uncontrolled hypertension
* Clinically significant abnormal findings on screening examination based on the Investigator's assessment
* Known hypersensitivity to clomiphene
* Symptomatic cataracts
* Presence or history of known hyperprolactinemia with or without a tumor
* End-stage renal disease
* Any contraindication to testosterone supplementation therapy
* Absolute contraindications to hormone supplementation therapy which include active prostate cancer (or suspicion of prostate disease unless ruled out by biopsy), prostatic specific antigen (PSA)>=3.6, breast cancer, hematocrit>=51% (hemoglobin>=17 g/dL), uncontrolled congestive heart failure (CHF), myocardial infarction, acute coronary event, unstable angina, coronary revascularization procedure in the preceding 6 months, untreated obstructive sleep apnea, high risk of prostate cancer (ethnicity or family history), or severe lower urinary tract symptoms (AUA symptom score>19).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter N Schlegel, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, Department of Urology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Weill Cornell Medical College, Department of Urology — http://www.cornellurology.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Clomiphene Citrate: The initial dose of clomiphene citrate will be 25 mg (po, pill by mouth) every other day. This will be started at visit 2, week 0 of the study following diagnosis of low baseline testosterone (serum total testosterone <350 ng/dl in men <55 years, <300 ng/dl in men 55-65 years). Clomiphene citrate dose will be titrated up to a maximum of 50 mg daily according to serum total testosterone levels measured at follow-up visits during the 3 month duration of the study.
  Clomiphene citrate
Period: Overall Study
Arm/Group | Clomiphene Citrate | Placebo
Started | 6 | 7
Completed | 5 | 6
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clomiphene Citrate | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 2 | 5 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Serum Total Testosterone (Change From Baseline)
Description: Morning venipuncture of serum total testosterone.
Time Frame: 3 months post initial visit
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Clomiphene Citrate | Placebo
Number analyzed (Participants) | 5 | 6
ng/mL | 322.5 (40.9) | 179.8 (72.2)

2. Secondary Outcome: Other Hormonal Profile (Change From Baseline)
Description: Luteinizing hormone (LH)
Time Frame: 3 months post initial visit
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Clomiphene Citrate | Placebo
Number analyzed (Participants) | 5 | 6
IU/mL | 3.3 (2.4) | 2.2 (1.2)

3. Secondary Outcome: Androgen Deficiency in the Aging Male (ADAM) Questionnaire
Description: Overall, study subjects will be assessed for possible change in hypogonadal, sexual function, and pain symptoms. Minimum score is 0 and maximum score is 10. 0 is most symptomatic, and 10 is least symptomatic.
Time Frame: 3 months post initial visit
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Clomiphene Citrate | Placebo
Number analyzed (Participants) | 5 | 6
scores on a scale | 8.0 (1.6) | 8.0 (2.1)

4. Secondary Outcome: Hematocrit (%)
Description: Measure hematocrit from baseline.
Time Frame: 3 months post initial visit
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Clomiphene Citrate | Placebo
Number analyzed (Participants) | 5 | 6
percentage | 35.2 (12.8) | 42.3 (3.5)

5. Secondary Outcome: Estradiol
Time Frame: 3 months post initial visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Clomiphene Citrate | Placebo
Number analyzed (Participants) | 5 | 6
pg/mL | 23 (4.1) | 25.2 (7.6)

6. Secondary Outcome: Sexual Health Inventory for Men (SHIM) Questionnaire
Description: Overall, study subjects will be assessed for possible change in hypogonadal, sexual function, and pain symptoms. Minimum score is 1, maximum score is 25. The minimum value is most symptomatic and maximum value is least symptomatic.
Time Frame: 3 months post initial visit
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Clomiphene Citrate | Placebo
Number analyzed (Participants) | 5 | 6
scores on a scale | 12.2 (4.0) | 18.5 (5.8)

7. Secondary Outcome: Men's Sexual Health Questionnaire (MSHQ) Questionnaire
Description: Overall, study subjects will be assessed for possible change in hypogonadal, sexual function, and pain symptoms. Minimum score is 1, maximum score is 20. Minimum score is considered most symptomatic, maximum score is considered least symptomatic.
Time Frame: 3 months post initial visit
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Clomiphene Citrate | Placebo
Number analyzed (Participants) | 5 | 6
scores on a scale | 7.0 (1.2) | 8.8 (4.3)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Clomiphene Citrate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes